CLINICAL TRIAL: NCT01372267
Title: Psychosocial Pain Management During Addictions Treatment to Improve Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Mark A. Ilgen, Associate Professor of Psychiatry, Medical School, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1R01DA029587-01A1 (NIH)
Record Dates: First submitted 2011-06-07; First posted 2011-06-13 (Estimated); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Pain
Keywords: Cognitive Behavioral Therapy; Chronic Pain; Substance Use Disorders; Psychoeducational control group
MeSH Terms: conditions — Pain; Chronic Pain; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT for pain (Experimental)
  Interventions: Behavioral: CBT for pain in Substance abuse
- Psychoeducational control group (Active Comparator): This group is designed to be an active control which provides detailed information about substance us and chronic pain without providing any CBT or other specific therapy.
  Interventions: Behavioral: Psychoeducation for substance abuse

INTERVENTIONS:
Behavioral: Psychoeducation for substance abuse — This active control provides detailed educational information about substance use and chronic pain to those enrolled.
  Arms: Psychoeducational control group
Behavioral: CBT for pain in Substance abuse — The therapeutic intervention group is designed to provide beneficial coping strategies that are helpful in dealing with both substance use and pain.
  Arms: CBT for pain

SUMMARY:
The present intervention is a Stage II randomized controlled efficacy trial of a group-based intervention that integrates Cognitive Behavioral Therapy (CBT) for pain and substance use disorders (SUDs) compared to a Supportive Psychoeducation Control (SPC) group in a sample of patients receiving residential SUD treatment with co-occurring chronic pain. A total of 452 patients (226 male and 226 female) with current pain rated as moderately severe or greater and comorbid drug or alcohol use disorder(s) will be recruited from a large residential SUD treatment program. These participants will be randomly assigned to either a 4-week (8-session) group of integrated CBT for pain and SUDs or a 4-week (8-session) SPC group. All participants will be re-assessed immediately post-treatment (1 month) and again at 3, 6, and 12 months post-intervention. Through this randomized controlled trial, the investigators hope to gain insight on how to improved treatment of pain in those with SUDs that could result in enhanced quality of life and improved pain-related, substance use, and other health outcomes. Evaluating a psychosocial intervention for pain and substance use that can be delivered during a SUD treatment episode would significantly extend available treatment options for the large numbers of patients with pain seen by SUD treatment providers. The investigators also hope to determine the efficacy of an evidence-based psychosocial pain management approach in men and women from a large and diverse residential addiction treatment program.

DETAILED DESCRIPTION:
Chronic pain among individuals who misuse drugs or alcohol is a common and critically important problem that is rarely managed appropriately. The estimated rates of chronic pain in Substance Use Disorder (SUD) treatment are as high as 60%. Chronic pain is seldom successfully addressed in SUD treatment settings because of a limited understanding of the problem and a lack of effective intervention strategies. A clear and urgent need exists for the study of effective alternatives to the use of opiate pain medications in those treated for SUDs who also have pain because of: (1) the potential for abuse and diversion of opiate medications by patients in SUD treatment; and (2) recent evidence that untreated pain may undermine the effectiveness of standard treatments for SUDs.

An important potential strategy to address this problem is the use of Cognitive Behavioral Therapy (CBT) to manage pain and decrease substance misuse. Psychosocial interventions such as CBT have demonstrated efficacy for reducing pain and improving functioning for a broad spectrum of pain-related conditions. However, this form of treatment has not been explicitly tested in patients with co-occurring substance use disorders. Additionally, although pain is common in both men and women, most studies have lacked sufficient power to test the effect of interventions separately in men and women. The present intervention is designed to integrate CBT for pain and CBT for SUDs with the primary goal of improving pain- and substance-related outcomes. The investigators will test the efficacy of this modified protocol on both men and women in this understudied patient population.

ELIGIBILITY:
Inclusion Criteria:

* Must be over 18 years of age
* Report moderate to severe pain over past 3 months
* Resided in treatment for less than 60 days

Exclusion Criteria:

* Acute suicidality
* Mental incompetence (e.g. unable to provide informed consent)
* Evidence of current psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510 (Actual)
Dates: Start 2011-10; Primary Completion 2016-01 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Change in level of pain | Baseline, one, three, six, twelve months
  For each follow-up time point, we will subtract the baseline value to obtain a change score
Change in pain tolerance | Baseline, one, three, six, twelve months
  For each follow-up time point, we will subtract the baseline value to obtain a change score
Change in pain-related functioning | Baseline, one, three, six, twelve months
  For each follow-up time point, we will subtract the baseline value to obtain a change score

SECONDARY OUTCOMES:
Change in Substance use | Baseline, three, six, twelve months

CONTACTS AND LOCATIONS:
Locations (1):
- Community Programs, INC., Waterford, Michigan, United States

REFERENCES:
- [Derived] Ilgen MA, Coughlin LN, Bohnert ASB, Chermack S, Price A, Kim HM, Jannausch M, Blow FC. Efficacy of a Psychosocial Pain Management Intervention for Men and Women With Substance Use Disorders and Chronic Pain: A Randomized Clinical Trial. JAMA Psychiatry. 2020 Dec 1;77(12):1225-1234. doi: 10.1001/jamapsychiatry.2020.2369. PMID 32725178